CLINICAL TRIAL: NCT01521975
Title: A Two-year, Open-label, Virological Response Adaptive Design, Multicenter Study to Evaluate Efficacy of Telbivudine in HBeAg Negative Adult CHB Patients With Roadmap Strategy
Brief Title: A Two-year Study of Telbivudine in HBeAg Negative Hepatitis
Acronym: STEN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Guangzhou 8th People's Hospital (Other)
Responsible Party: Principal Investigator, Chao-Shuang Lin, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBeAg negative Roadmap
Record Dates: First submitted 2012-01-26; First posted 2012-01-31 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2011-01

CONDITIONS: Hepatitis B, Chronic
Keywords: HBV DNA; LdT; ADV; HBeAg negative hepatitis; CHB
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine; adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HBeAg Negative Hepatitis (Experimental): HBeAg Negative Hepatitis patients.
  Interventions: Drug: Telbivudine, Adefovir dipivoxil

INTERVENTIONS:
Drug: Telbivudine, Adefovir dipivoxil — All patients will take Telbivudine 600 mg PO daily from baseline. Some patients will take Adefovir dipivoxil 10 mg PO daily if they meet the criteria of adding Adefovir dipivoxil.
  Other Names: Sebivo, LDT

SUMMARY:
Based on GLOBE study supplying predictability analysis results, ROADMAP strategy provides an individualized telbivudine treatment roadmap strategy designed to achieve optimal viral suppression and low resistance rate in patients with chronic hepatitis B(CHB), which includes adding ADV treatment at different time points according to individual patient response. China CHB Guidelines (China Medical Association 2010) make impress on and confirm LDT ROADMAP strategy particularly, which may be a large potential to expand the naïve patients. We are lack of optimal model in HBeAg(-). In China HBeAg(-) is around 38% of total CHB patients. In GLOBE study, LdT treatment against HBeAg(-) patients with HBV DNA <7log showed a good 2 year efficacy, but we still look forward to more efficient treatment and lower resistance rate. This study complies with the principle of individualized therapy recommended and ethical principles. It is expected that this study design with individualized treatment approach may improve efficacy and lower the resistance rates. In addition, it will provide important information on how to bring greater benefits to patients with CHB.

DETAILED DESCRIPTION:
This study is an open-label, multicenter, PCR response adaptive clinical study design, with intensification of treatment (addition of adefovir to telbivudine treatment) depending on HBV DNA level at week 24. All patients commence with Telbivudine 600mg daily. At week 24 they will be divided into 2 Groups according to virological response. Patients with PCR detectable HBV DNA will add on ADV(Group I). Patients with PCR undetectable HBV DNA(Group II)will continue telbivudine monotherapy. ADV will not be added on unless viral breakthrough occurs.

ELIGIBILITY:
Inclusion Criteria:

* Detectable serum HBsAg at the Screening visit and at least 6 months prior
* HBeAg negative at Screening visit
* serum HBV DNA level >2,000 IU/mL at Screening visit
* Elevated serum ALT≥2 ×ULN and <10×ULN at Screening visit (excluding ALT elevations due to non-HBV reasons such as drug, alcohol etc)

Exclusion Criteria:

* Patient has a history of clinical signs/symptoms of hepatic decompensation (Child-Pugh Grade B or C) or ascites, esophageal variceal bleeding, hepatic encephalopathy, or spontaneous bacterial peritonitis.
* Patient has a history of hepatocellular carcinoma (HCC) or suspected symptoms of HCC, such as suspicious foci on imaging studies and/or serum alpha-fetoprotein (AFP)>50ng/mL.
* Patient has received treatment of nucleoside or nucleotide drugs whether approved or investigational before.
* Patient has received IFN or other immunomodulatory treatment within 52 weeks before Screening.
* Patient has a medical condition that requires frequent use of systemic acyclovir or famciclovir.
* Patient has a medical condition that requires frequent use of systemic corticosteroids, however topical and inhaled corticosteroids are allowed.
* Patient has used hepatotoxic drugs within one month.
* Patient has overtaken alcohol (>40g/day) or abused illicit drugs in recent one year.
* Use of other investigational drugs at the time of enrollment.
* History of hypersensitivity to any of the study drugs (telbivudine or adefovir).
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive urine pregnancy test.
* Patient is co-infected with HCV, HDV or HIV.
* Patient has one or more additional known primary or secondary causes of liver disease, other than hepatitis B (e.g., alcoholism, autoimmune hepatitis).
* History of malignancy of any organ system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2014-05-30 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with undectable HBV DNA | at Week 104

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Liang Gao, Prof, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Gan W, Li J, Zhang C, Chen X, Lin C, Gao Z. Efficacy of 104-week Telbivudine-based optimization strategy in patients with HBeAg-negative chronic hepatitis B virus infections. BMC Infect Dis. 2020 Dec 7;20(1):931. doi: 10.1186/s12879-020-05642-y. PMID 33287722